CLINICAL TRIAL: NCT02284412
Title: Visualization of Regional Lung Ventilation During Neostigmine or Sugammadex Enhanced Recovery From Moderate Residual Neuromuscular Blockade in the Anaesthetized Rat Using Functional Respiratory Imaging
Brief Title: Functional Respiratory Imaging After Neostigmine or Sugammadex
Acronym: FRINeoS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: Universiteit Antwerpen (Other); MSD Belgium BVBA (Industry)
Responsible Party: Principal Investigator, Guy CAMMU, MD, PhD, Onze Lieve Vrouw Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSGC02
Record Dates: First submitted 2014-10-28; First posted 2014-11-06 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Respiratory-Gated Imaging Techniques
Keywords: Neostigmine; Sugammadex
MeSH Terms: interventions — Neostigmine; Sugammadex; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- neostigmine (Active Comparator): Neostigmine will be dosed as 60 μg/kg, and glycopyrrolate 12 μg/kg (commercially available 5:1 co-formulation), as a single iv bolus administered over 10sec, for reversal of rocuronium-induced moderate neuromuscular blockade.
  Interventions: Drug: Neostigmine
- Sugammadex (Experimental): Sugammadex will be dosed 15 mg/kg, as a single iv bolus administered over 10sec, for reversal of rocuronium-induced moderate neuromuscular blockade.
  Interventions: Drug: Sugammadex
- Water for injection (Placebo Comparator): Water will be dosed arbitrarily as a 1 mL single iv bolus administered over 10sec.
  Interventions: Drug: Water for injection

INTERVENTIONS:
Drug: Neostigmine — At a train-of-four (TOF) ratio of 0.5: administration of neostigmine 0.06 mg/kg for reversal of neuromuscular blockade.
  Other Names: Robinul-Neostigmine
  Arms: neostigmine
Drug: Sugammadex — At a train-of-four (TOF) ratio of 0.5: administration of sugammadex 15 mg/kg for reversal of neuromuscular blockade.
  Other Names: Bridion
  Arms: Sugammadex
Drug: Water for injection — At a train-of-four (TOF) ratio of 0.5: administration of placebo for spontaneous recovery of neuromuscular blockade.
  Other Names: Aqua ad iniectabilia
  Arms: Water for injection

SUMMARY:
The use of neuromuscular blocking agents (NMBAs) is still associated with postoperative pulmonary complications. The investigators rely on acceleromyography (AMG) of a peripheral nerve/muscle to assess the patients' breathing capability at the end of surgery. It is possible that respiratory complications after surgery (e.g. desaturation and atelectasis) are related to the lack of diaphragm activity.

A previous trial by our study group links the use of sugammadex, a novel selective relaxant binding agent (SRBA) for reversal of neuromuscular blockade, to an increase in diaphragm electrical activity, compared to reversal with neostigmine. Our hypothesis is that by making nicotinergic acetylcholine receptors free from rocuronium in the diaphragmatic neuromuscular junctions, instead of increasing the amount of acetylcholine (like neostigmine does), sugammadex will result in a better neuromuscular coupling. This may have its subsequent effects on the central control of breathing, influencing the balance between intercostal and diaphragm activity.

The investigators now propose a study in rats, where the investigators will use Functional Respiratory Imaging (FRI, property of FluidDA n.v., Groeningenlei 132, B-2550 Kontich) to assess regional lung ventilation after sugammadex, neostigmine or spontaneous reversal. The images obtained through micro-CT scans allow us to accurately reconstruct airway morphology in the free-breathing rat. It will provide us with new insights into breathing physiology after reversal of neuromuscular blockade.

DETAILED DESCRIPTION:
This study is designed to assess the effect of sugammadex, neostigmine/glycopyrrolate and spontaneous reversal of a moderate rocuronium-induced neuromuscular blockade on regional lung ventilation. This is a randomized, controlled, parallel-group double blind trial in rats. A total of 18 adult male Sprague-Dawley rats will be used, 6 in each treatment group. The animals will be randomized in one of three groups, in a 1:1:1 ratio. This randomization will be performed according to a computer-generated randomization list. The first group will receive neostigmine/glycopyrrolate. The second group will receive sugammadex. The third group will receive water for injection. Reversal agents will be administered at a train-of-four (TOF) of 0.5, as measured with AMG.

The investigators will assess regional ventilation by means of micro-CT scanning during spontaneous breathing after the TOF ratio has reached ≥ 0.9. This way, the investigators can accurately reconstruct airway morphology. The different airway sections can then be linked to the corresponding lung tissue, and a full anatomical picture is thus rendered. A comparison of morphological scans at different breathing levels (e.g. end-inspiratory and end-expiratory) will allow us to model breath-by-breath regional airway and alveolar recruitment.

ELIGIBILITY:
Inclusion Criteria:

* male Sprague-Dawley rats

Exclusion Criteria:

* N/A

Ages: 3 Months to 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Regional lung ventilation assessed by means of micro-CT scanning during spontaneous breathing after recovery from neuromuscular block. | CT scanning will take between 5 to 8 minutes, followed by post-processing of the images.
  Comparison of the effect of sugammadex, neostigmine/glycopyrrolate and spontaneous recovery on regional lung ventilation in the spontaneously breathing rat, assessed by micro-CT scanning after recovery from neuromuscular block.

SECONDARY OUTCOMES:
Tidal volume (TV, mL) of breaths recorded by means of micro-CT scanning during spontaneous breathing after recovery from neuromuscular block. | CT scanning will take between 5 to 8 minutes, followed by post-processing of the images.
  Comparison of the effect of sugammadex, neostigmine/glycopyrrolate and spontaneous recovery on tidal volume of breaths in the spontaneously breathing rat, assessed by micro-CT scanning after recovery from neuromuscular block.

CONTACTS AND LOCATIONS:
Overall Officials: GUY CAMMU, MD, PhD, Principal Investigator — OLV Hospital, Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

REFERENCES:
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Cammu GV, Smet V, De Jongh K, Vandeput D. A prospective, observational study comparing postoperative residual curarisation and early adverse respiratory events in patients reversed with neostigmine or sugammadex or after apparent spontaneous recovery. Anaesth Intensive Care. 2012 Nov;40(6):999-1006. doi: 10.1177/0310057X1204000611. PMID 23194209
- [Background] Grosse-Sundrup M, Henneman JP, Sandberg WS, Bateman BT, Uribe JV, Nguyen NT, Ehrenfeld JM, Martinez EA, Kurth T, Eikermann M. Intermediate acting non-depolarizing neuromuscular blocking agents and risk of postoperative respiratory complications: prospective propensity score matched cohort study. BMJ. 2012 Oct 15;345:e6329. doi: 10.1136/bmj.e6329. PMID 23077290
- [Background] Schepens T, Cammu G, Saldien V, De Neve N, Jorens PG, Foubert L, Vercauteren M. Electromyographic activity of the diaphragm during neostigmine or sugammadex-enhanced recovery after neuromuscular blockade with rocuronium: a randomised controlled study in healthy volunteers. Eur J Anaesthesiol. 2015 Jan;32(1):49-57. doi: 10.1097/EJA.0000000000000140. PMID 25111539
- [Background] De Backer JW, Vos WG, Burnell P, Verhulst SL, Salmon P, De Clerck N, De Backer W. Study of the variability in upper and lower airway morphology in Sprague-Dawley rats using modern micro-CT scan-based segmentation techniques. Anat Rec (Hoboken). 2009 May;292(5):720-7. doi: 10.1002/ar.20877. PMID 19322825
- [Background] Eikermann M, Zaremba S, Malhotra A, Jordan AS, Rosow C, Chamberlin NL. Neostigmine but not sugammadex impairs upper airway dilator muscle activity and breathing. Br J Anaesth. 2008 Sep;101(3):344-9. doi: 10.1093/bja/aen176. Epub 2008 Jun 16. PMID 18559352